CLINICAL TRIAL: NCT03660670
Title: Medico-economic Evaluation of the ONCORAL Program of Multidisciplinary ONCOlogic Interventions Between Town and Hospital (Doctor-pharmacist-nurse) for Ambulatory Patients Under oRAL Anticancer Drugs Versus Usual Care
Brief Title: Medico-economic Evaluation of the ONCORAL Program for Ambulatory Patients Under Oral Anticancer Drugs Versus Usual Care
Acronym: ONCORAL-PRME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL18_0046
Record Dates: First submitted 2018-08-16; First posted 2018-09-06 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: Oral chemotherapy; cancer outpatient; ONCORAL; medico-economic; Health related program; multidisciplinary; therapeutic education
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm (Experimental): Application of the ONCORAL program of multidisciplinary ONCOlogic interventions between town and hospital (doctor-pharmacist-nurse) for ambulatory patients under oRAL anticancer drugs
  Interventions: Behavioral: ONCORAL therapeutic education
- Standard of care (Sham Comparator): Patients in the control group will receive regular follow-up from their oncologist, but no more that the standard care.
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: ONCORAL therapeutic education — Multidisciplinary program that includes informative cessions with a hospital pharmacist about the anticancer drug: information is given to the patients on adverse events and their managements, optimizing drug dosage plans. Moreover, information is shared with town partners: doctor, pharmacists, and nurses.
  Arms: Interventional Arm
Behavioral: Standard of care — In the group of standard of care, patients will have interviews with a clinical research associate only dedicated to the record of data for outcomes assessments.
  Arms: Standard of care

SUMMARY:
Economic impact of cancer treatments is increasing for years: increase of number of patients (385 000 new occurrences in 2015), increase of life expectancies, chronicization of diseases and increase of therapeutic innovation costs.

Oral anticancer drugs allow the ambulatory turn in oncologic treatments, avoid hospitalizations dues to injectable chemotherapies and improve patient autonomy. In real life situation, these drugs still remain linked to significant drug iatrogenic effects: prevalent adverse events and potentially serious ones, drugs interactions for one other patient, considered as major in 15-20% cases, and non-observance for 30-50% patients.

The resultant care overconsumption and the high cost of new oral targeted therapies appear as a substantial financial charge to the Health related program. Securing oral chemotherapy and their good practice therefore represent a real economic challenge and lead health care professionals to develop town-hospital programs of ambulatory patient's follow-up under oral anticancer drug in response of third Cancer Plan.

Benefice of such interventions are proved on observance, management of adverse events and drug interactions.

However, the effectiveness of these programs has not been evaluated and no studies have been conducted in France.

The Investigators propose here to carry out a medico-economic study of high level of proof of the ONCORAL program. This study will be the first evaluation of the effectiveness of a program for monitoring outpatient oral cancer patients versus usual care.

The results of this study will contribute to the national reflection on the path of care of patients treated by oral chemotherapy, on the assessment of needs and the evolution of the supply of care and its financing.

ELIGIBILITY:
Inclusion Criteria:

* Adult more than 18 years-old
* Cancer patient
* For whom an initiation or a change of oral anticancer is prescribed according to the AMM
* Considered by the oncologist as at iatrogenic drug risk, or having 3 or more risk factors, to develop an iatrogenic drug issue among the following risk factors:
* ≥ 2 oral anticancer drugs,
* ≥ 2 lines of treatment,
* combination with an injectable chemotherapy,
* rhythm discontinuous intake of oral anticancer,
* ≥ 2 associated chronic conditions,
* number of associated drugs including oral anticancer ≥5,
* creatinine clearance <60 ml / min,
* frailties and psychosocial conditions at risk (isolated patient, foreign, having limited autonomy)
* without major psychiatric cognitive impairment that may interfere with the ONCORAL program;
* in sufficient autonomy to manage his home treatment;
* signed a written informed consent to participate;
* Affiliate or beneficiary of a Social Security or similar.

Exclusion Criteria:

* Treated with oral anticancer in a clinical trial or temporal use authorization
* Management of oral anticancer treatment exclusively by the caregiver;
* Who did not report a regular physician or pharmacy, or who reported ≥2 or more regular street pharmacies;
* In an institution or guardianship, a major protected by the law;
* Participation in a clinical trial that may alter the costs of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate efficiency of ONCORAL program for ambulatory patients under oral anticancer drugs versus usual care | Month 12
  Efficiency is calculated on the double dimension cost and year of life corrected by quality of life (QALY).

SECONDARY OUTCOMES:
Evaluate the cost price in charge for the two strategies | Month 12
  Medico-economic datas will be assessed in parallel of the clinical study. All costs for Health related program will be added during 12 months : nonscheduled hospitalizations due to drugs issues, medical consultations, time spent by the hospital pharmacist, time spent by the nurse, time spent with town partners sharing information, biological or radiological exams done, nursing in town or at home.
Patient's quality of life, measured with the EQ-5D-3L (EuroQol Group-5 dimensions-3 levels) questionnaire | at inclusion, 3 months, 6 months and 12 months post inclusion
  The questionnaire is a descriptive system comprises five dimensions. Each dimension has 3 levels : no problems, some problems, and extreme problems. EQ-5D health states, may be converted into a single summary index by applying a formula that essentially attaches values (also called weights) to each of the levels in each dimension. The averages of the EQ-5D-3L scores, summarized and for each sub-dimension, will be calculated in each group at baseline, 3 months, 6 months, and 12 months post-inclusion.
Budget impact analysis of 12-months of ONCORAL care. | 12 months
  Costs of the introduction of ONCORAL program on the Health Insurance budget.
Oral anti-cancer dose taken relative to the dose of the marketing authorization | 3, 6 and 12 months post-inclusion
  For each patient, the number of oral anti-cancer units really taken by the patient will be calculated from the data obtained by the delivery of treatments (and reported units) in city pharmacy or retrocession. This number will be compared to the total number of units that should have been taken if he had received the treatment in accordance with the marketing authorization of the oral anticancer drug. In each group and for each time, the averages, standard deviations, and quartiles observed in each arm will be calculated.
Reasons for modifications of relative dose-intensity | 3, 6 and 12 months post-inclusion
  For each patient, the number of oral anti-cancer units actually taken by the patient will be calculated from the data from the delivery of treatments in town pharmacy or retrocession and reported units. This number will be related to the total number of units that should have been taken if he had received the treatment in accordance with the AMM of the oral anticancer drug. For each reason type of changes in relative dose-intensity, and for the causes of the changes, the proportions observed in each of the groups will be calculated
Observance of oral anti-cancer drugs | 3, 6 and 12 months post-inclusion
  Adherence will be measured with a 6-item medication adherence scale (adherence will be defined as a score ≤ 2) and the rate of prescription renewal by the ambulatory pharmacy (adherence will be defined as a rate ≥80%).
Adverse events related to oral anti-cancer drug | From baseline to 12 months
  For each type of adverse event related to SOC oral anticancer, and for each CTCAE grade, the proportions observed in each group will be calculated between baseline and 12 months. The clinical consequences according to the NCCMERP scale will be described; their proportions will be calculated for each group.
Drug interactions | From baseline to 12 months
  For each type of drug interaction (contraindication, not recommended association, precaution of use) related to the oral anticancer drug between the inclusion and 12 months, the proportions observed in each of the groups will be calculated. The clinical consequences according to the DDI Predictor software will be described.
Medication errors | From baseline to 12 months
  For each type of drug error confirmed and related to the oral anticancer drug between baseline and 12 months, the proportions observed in each group will be calculated. The clinical consequences according to the NCCMERP scale will be described; their proportions will be calculated for each group.
Overal survival evaluation | 12 months
  The overall survival rate of the disease will be estimated up to 12 months post-inclusion using a Kaplan-Meier model. A Log-rank test will be implemented to compare overall survival rates between the two groups.
Progression free survival evaluation | 12 months
  The progression-free survival rate of the disease will be estimated up to 12 months post-inclusion using a Kaplan-Meier model. A Log-rank test will be implemented to compare progression free survival rates between the two groups.
Patient Satisfaction Score for Therapeutic care | 3, 6, 9 and 12 months
  The mean scores in SAT-MED Q (Treatment Satisfaction with Medicines Questionnaire) scale will be calculated for each of the two groups. The Sat-Med Q is a self-questionnaire of seventeen questions grouped into six elements; effectiveness, side effects, comfort of use, the general opinion of the patient, evaluation of the effect of the treatment on the patient's daily life, as well as the quality of the follow-up and the information provided by the patients. The answers are expressed on a scale of 5 points. from "No, not at all = 0 points" to "Yes, many = 4 points". Totaling the direct scores of the items yields a total composite score ranging between 0 and 68. The resultant total composite score can be transformed to a more intuitive and easier to understand metric with a minimum of 0 and a maximum of 100, using a mathematic expression.
Disease representation from patient | baseline, 6 months and 12 months
  The mean total scores and in each dimension of the B-IPQ (Brief Illness Perception Questionnaire) scale will be calculated for each of the two groups. The Brief IPQ has nine items. All of the items except the causal question are rated using a 0-to- 10 response scale. Five of the items assess cognitive illness representations, two of the items assess emotional representations and one item assesses illness comprehensibility. Assessment of the causal representation is by an openended response item. A mixed repeated measures model will be realized to estimate its evolution. The link between variation in disease representations between inclusion and final assessment and adherence, dose-relative intensity, and quality of life will be tested using a multivariate linear regression model.
Treatment representation from patient's point of view | baseline, 6 months and 12 months
  The total average scores of the BMQ scale will be calculated in each dimension for each of the two groups. A mixed repeated measures model will be realized to estimate its evolution. The relationship between variation in treatment representations and adherence, dose-relative intensity, and quality of life between inclusion and final assessment will be tested using a multivariate linear regression model.
Perceived social support | 6 and 12 months
  This criterion is in the form of 4-level Likert scales, concerning 3 items (support of the person with whom the patient lives in a couple, support of family members, support of friends and relatives), and for each two-dimensional item (psychological support and material support). Each dimension of each item will be analyzed independently. At each measurement, the response will be compared to that given during the previous visit. A break in perceived support will be considered if the response goes from 3 "a lot" to 0 "not at all", 1 "a little" or 2 "moderately". At each time, the percentage of patients with perceived support disruption will be calculated for each item and dimension, in each of the two groups, and these percentages will be compared. An analysis of the factors influencing the occurrence of perceived support disruption will be performed using a multivariate linear regression model.
Health locus of control of the patient | baseline, 6 months and 12 months post-inclusion
  The average scores on the Doran TSCT scale will be calculated in each group. A mixed repeated measures model will be realized to estimate its evolution. The link between self-management variation (TSCT score) and adherence, dose-relative intensity, and quality of life between inclusion and final assessment will be tested using a linear regression multivariate model.
Quality of life of patients | baseline, 3 months, 6 months, and 12 months post-inclusion
  The averages of the QLQ-C30 scores, summarized and for each sub-dimension, will be calculated in each group. A mixed repeated-measures model will be constructed to estimate the evolution of quality of life over time and compare it between the two groups.
For investigational arm : patient's reported adverse events | From baseline to 12 months
  A description of the number, the percentages according to the Standard Of Care, and a list of the modalities of management of the adverse events grades 2, 3 and 4 reported by the patient in his city-hospital liaison booklet related to the oral anticancer drug will be performed.
Satisfaction of first resort (doctor, pharmacist and liberal nurse) | 12 months
  The averages, standard deviations, and quartiles observed will be calculated for each category of interviewee on his satisfaction with the ONCORAL program (with the use of a visual analogic scale EVA, from 0 to 10).
Satisfaction of patient | 12 months
  The averages, standard deviations, and quartiles observed will be calculated for the patient on his satisfaction with the ONCORAL program (with the use of a visual analogic scale EVA, from 0 to 10).
Types of pharmaceutical interventions | 12 months
  Number and types of pharmaceutical interventions as part of the city-hospital link according to the ACT-IP score adaptation during the 12-month post-inclusion period

CONTACTS AND LOCATIONS:
Overall Officials: Catherine RIOUFOL, PharmD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No
Sharing of individual data have not been planned

REFERENCES:
- [Derived] Huot L, Guerre P, Descotes G, Caffin AG, Herledan C, Ranchon F, Rioufol C. Cost-effectiveness of the ONCORAL multidisciplinary programme for the management of outpatients taking oral anticancer agents at risk of drug-related event: protocol for a pragmatic randomised controlled study. BMJ Open. 2024 Feb 17;14(2):e074956. doi: 10.1136/bmjopen-2023-074956. PMID 38367968